CLINICAL TRIAL: NCT01433497
Title: A 96 Week, Prospective, Multicentre, Randomized, Double-blind, Placebo-controlled, 2 Parallel-groups, Phase 3 Study to Compare Efficacy and Safety of Masitinib 4.5 mg/kg/Day Versus Placebo in the Treatment of Patients With Primary Progressive or Relapse-free Secondary Progressive Multiple Sclerosis
Brief Title: Efficacy and Safety of Masitinib in the Treatment of Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB07002
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Relapse Free
Keywords: multiple sclerosis; primary progressive; relapse-free; secondary progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Experimental Arm A (Experimental): Participants receive masitinib (4.5 mg/kg/day), given orally twice daily.
  Interventions: Drug: Masitinib
- Experimental Arm B (Experimental): Participants receive masitinib (4.5 mg/kg/day), given orally twice daily, with a dose escalation to 6 mg/kg/day after 3 months of treatment.
  Interventions: Drug: Masitinib
- Placebo Comparator A (Placebo Comparator): Participants receive placebo given orally twice daily.
  Interventions: Drug: Placebo
- Placebo Comparator B (Placebo Comparator): Participants receive placebo, given orally twice daily, with a matched dose escalation after 3 months of treatment.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Masitinib
  Other Names: AB1010
  Arms: Experimental Arm A; Experimental Arm B
Drug: Placebo
  Other Names: Placebo Oral Tablet
  Arms: Placebo Comparator A; Placebo Comparator B

SUMMARY:
The purpose of this study is to compare the safety and efficacy of masitinib 6 mg/kg/day versus placebo in the treatment of patients with primary progressive multiple sclerosis or relapse-free secondary progressive multiple sclerosis.

DETAILED DESCRIPTION:
Masitinib is a selective tyrosine kinase inhibitor that is thought to exert a neuroprotective effect through its activity on mast cells and other non-neuronal cells of the central nervous system, with subsequent modulation of inflammatory and neurodegenerative processes. The objective of this study is to compare the efficacy and safety of masitinib at 4.5 mg/kg/day versus matched placebo, or masitinib at 4.5 mg/kg/day with a dose escalation to 6 mg/kg/day after 3 months of treatment versus matched placebo, in the treatment of patients with primary progressive multiple sclerosis or relapse-free secondary progressive multiple sclerosis. Approximately 600 patients will be randomized into four treatment groups with a 2:2:1:1 design. The primary outcome measure is the Expanded Disability Status Scale (EDSS) after 96 weeks of treatment in the overall study population with subgroup analysis performed in stratum (primary progressive multiple sclerosis / secondary progressive multiple sclerosis).

ELIGIBILITY:
Main inclusion criteria:

- Patient suffering from either primary progressive or secondary progressive multiple sclerosis without relapse within 2 years before inclusion according to the revised McDonald's criteria.

Main exclusion criteria:

- Patient suffering from a disease other than MS that would better explain the patient's neurological clinical signs and symptoms and/or MRI lesions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
EDSS | 96 weeks
  Expanded Disability Status Scale (EDSS) after 96 weeks of treatment

SECONDARY OUTCOMES:
MSQOL-54 | 96 weeks
  Multiple Sclerosis Quality of Life 54 items (MSQOL-54)
MSFC | 96 weeks
  Multiple Sclerosis Functional Composite (MSFC)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Vermersch, MD, PhD, Principal Investigator — Hôpital Salengro, Lille, France
Locations (8):
- "St. Ivan Rilski" University Multiprofile Hospital for Active Treatment, Sofia, Bulgaria
- France (2):
  - GHICL hopital ST vincent de Paul, Lille
  - Hôpital de Gui de Chauliac, Montpellier
- Universitätsklinikum Gießen und Marburg, Marburg, Germany
- Rehibilitation Center "KENTAVROS", Volos, Greece
- KO-MED Centra Kliniczne Lublin II, Lublin, Poland
- Centrul Medical Clubul Sănătăţii, Campulung Muscel, Romania
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

REFERENCES:
- [Derived] Vermersch P, Brieva-Ruiz L, Fox RJ, Paul F, Ramio-Torrenta L, Schwab M, Moussy A, Mansfield C, Hermine O, Maciejowski M; AB07002 Study Group. Efficacy and Safety of Masitinib in Progressive Forms of Multiple Sclerosis: A Randomized, Phase 3, Clinical Trial. Neurol Neuroimmunol Neuroinflamm. 2022 Feb 21;9(3):e1148. doi: 10.1212/NXI.0000000000001148. Print 2022 May. PMID 35190477